CLINICAL TRIAL: NCT02462044
Title: Contrast Enhancement on Coronary Computed Tomographic Angiography : Effects on Intra-Coronary Attenuation Using Low Iodine Concentrations While Maintaining Identical IDR (EICAR-Trial)
Brief Title: Contrast Enhancement on Coronary Computed Tomographic Angiography
Acronym: EICAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Marco Das, Marco Das, MD, PhD, Maastricht University Medical Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: METC 13-1-033
Record Dates: First submitted 2014-09-09; First posted 2015-06-03 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Coronary Artery Disease; Coronary Stenosis
Keywords: Computed tomography; Coronary CTA; Contrast media
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis | interventions — Iodine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 240 (Experimental): Group 240 will receive CM with 240 mg Iodine/ml IDR 2.0 gI/s
  Interventions: Drug: 240 mg Iodine
- 300 (Experimental): Group 300 will receive CM with 300 mg Iodine/ml IDR 2.0 gI/s
  Interventions: Drug: 300 mg Iodine
- 370 (Experimental): Group 370 will receive CM with 370 mg Iodine/ml IDR 2.0 gI/s
  Interventions: Drug: 370 mg Iodine

INTERVENTIONS:
Drug: 240 mg Iodine
  Other Names: 240 mg Iodine/ml IDR 2.0 gI/s
  Arms: 240
Drug: 300 mg Iodine
  Other Names: 300 mg Iodine/ml IDR 2.0 gI/s
  Arms: 300
Drug: 370 mg Iodine
  Other Names: 240 mg Iodine/ml IDR 2.0 gI/s
  Arms: 370

SUMMARY:
Computed tomographic angiography (CTA) is an important prognostic tool with regard to the detection of coronary artery stenoses. Both iodine delivery rate (IDR; the amount of iodine delivered to the patient per second) and iodine concentration are decisive factors in the opacification of arterial vessels.

There remains to be some debate in the literature about whether the use of high iodine concentration contrast media is beneficial compared to lower iodine concentrations.

To date, there have not been any studies comparing intracoronary attenuation using concentrated contrast media lower than 300 mg I/ml at coronary CTA. For a reliable comparison of CM with different iodine concentrations, adapted injection protocols insuring an identical IDR (in g iodine per second) are mandatory. The investigators hypothesize that usage of lower iodine concentrations, while maintaining identical IDR and total iodine load, will result in comparable diagnostical intra-vascular attenuation in CTA.

DETAILED DESCRIPTION:
To evaluate intravascular contrast enhancement and image quality in coronary CTA using different iodine concentrations ranging from 240 to 370 mg iodine per ml, administered with an identical IDR and total iodine load.

To describe the effect of iodine concentration and flow rates on contrast bolus characteristics, eg time to peak, bolus homogeneity, injection pressure and patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Atypical or typical chest pain

Exclusion Criteria:

* Unstable angina
* Hemodynamic instability
* History of CAD
* Pregnancy
* Renal insufficiency (defined as glomerular filtration rate (GFR) <45ml/min or <60ml +diabetes
* HR > 90 bpm and the inability to receive beta-blockers and iodine allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
intravascular contrast enhancement | two years
  intravascular contrast enhancement and image quality based on different contrast media (240, 300, 370) as measured by circular ROI in the target vessels using dedicated post processing.

SECONDARY OUTCOMES:
time to peak | two years
  Effect of iodine concentration - as measured by dedicated contrast monitoring software.
bolus homogeneity | two years
  Effect on contrast bolus characteristics and injection pressure - as measured by dedicated contrast monitoring software.
patient comfort | two years
  Effect on patient comfort. As assessed by patient questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands